CLINICAL TRIAL: NCT01544556
Title: Use of PrineoTM (Dermabond Protape) Skin Adhesive for Wound Closure Following Abdominoplasty: An Open, Prospective, Controlled, Randomized Clinical Study
Brief Title: Use of PrineoTM (Dermabond Protape) Skin Adhesive for Wound Closure Following Abdominoplasty
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Daryousch Parvizi, MD, Resident, Medical University of Graz
Other Study IDs: Prineo 1; Prineo2 (Other: MUGraz)
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-02

CONDITIONS: Late Effects of Open Wound
Keywords: abdominoplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Prineo: An open, prospective, controlled, randomized clinical Study
- Steristrips: An open, prospective, controlled, randomized clinical Study

SUMMARY:
Abdominoplasty is one of the most commonly performed procedures in plastic surgery. The appearance of the scar is a major factor contributing to the aesthetic outcome of the procedure and depends largely on the technique of wound closure. The investigators routinely used resorbable subcutaneous sutures and resorbable intracutaneous sutures for this closure. To overcome the potential detrimental effects of sutures in skin closure, surgical adhesives were introduced as a new technology. The new PrineoTM wound closure system was created to combine the effectiveness of 2-octyl-cyanoacrylate (Dermabond TM) together with a self-adhering mesh to make closure of long skin incisions even more safe and reliable. PrineoTM has the potential to offer a patient several benefits over traditional wound closure with sutures.A patient treated with Prineo™ can shower immediately following a procedure because the product forms a watertight barrier over the incision. PrineoTM can be easily removed, often with less pain than is sometimes associated with suture removal, after the natural wound healing process is complete (approximately 12 to 25 days). Other benefits are that it forms a microbial barrier and provides even distribution of tension across the length of the incision to ensure wound edge approximation throughout the wound healing process. Furthermore, it reduces subcuticular closure time as compared to subcuticular suturing.

However, these potential advantages have not been proven until now, as the methods used to assess the aesthetic outcome were not reproducible in most assessments, and none of these studies assessed patient satisfaction.1-3 Moreover, none was performed in a plastic surgical patient population. For these reasons, the investigators prospectively studied the results of wound closure after abdominoplasty with randomized use of PrineoTM and conventional suturing to assess the possible difference in outcome between these two methods.

DETAILED DESCRIPTION:
Abdominoplasty is one of the most commonly performed procedures in plastic surgery. The appearance of the scar is a major factor contributing to the aesthetic outcome of the procedure and depends largely on the technique of wound closure. The new PrineoTM wound closure system was introduced to combine the effectiveness of 2-octyl-cyanoacrylate (Dermabond TM) together with a self-adhering mesh.Fifty-two women and 8 men aged between 21 and 65 years scheduled for abdominoplasty were included in the study. Two weeks postoperatively, the wounds were examined and graded according to the Hollander Cosmesis Scale. At 3- and 6-month follow-up, the aesthetic outcome of the abdominal scar was evaluated with the Vancouver Scar Scale. Six months postoperatively, the patients were further asked to score their part of the Patient Scar Assessment Scale.The Hollander Cosmesis Scale indicated a significantly more favourable overall result with PrineoTM at 2 weeks after surgery. The Vancouver Scar Scale demonstrated a better cosmetic outcome in favour of PrineoTM 3 and 6 months after surgery The Patient Scar Assessment Scale scores 6 months after surgery indicated that the patients noted significantly less pain, thickness and irregularity with PrineoTM.Based on the investigators results, the investigators conclude that PrineoTM is a safe and effective substitute for superficial skin closure, with good cosmetic results and no increase in wound complications. The use of PrineoTM decreases operative times and enhances patients' postoperative comfort

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

peripheral vascular disease; insulin dependent diabetes mellitus; current intake of systemic steroids; known HIV-positive or other immunocompromised status; known or suspected allergy or sensitivity to cyanoacrylate, formaldehyde, tapes or adhesives; personal or family history of keloid or hypertrophic scar formation; or additional surgical procedures performed in the same surgical session in the same anatomical region. -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty-two women and 8 men aged between 21 and 65 years scheduled for abdominoplasty were included in the study.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2009-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Plastic, Aesthetic and Reconstructive Surgery, Department of Surgery,Medical University of Graz, Austria, Graz, Styria, Austria